CLINICAL TRIAL: NCT04283461
Title: Phase I, Open-Label, Dose-Ranging Study of the Safety and Immunogenicity of 2019-nCoV Vaccine (mRNA-1273) in Healthy Adults
Brief Title: Safety and Immunogenicity Study of 2019-nCoV Vaccine (mRNA-1273) for Prophylaxis of SARS-CoV-2 Infection (COVID-19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 20-0003; 5UM1AI148373-05 (NIH)
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2021-08-26

CONDITIONS: COVID-19; COVID-19 Immunisation
Keywords: 2019-nCoV (mRNA-1273); COVID-19; Dose-escalation; Immunogenicity; novel coronavirus; Safety; SARS-CoV-2; vaccine
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- Arm 1 (Experimental): 25 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age. N=15 (4 sentinel, 11 non-sentinel)
  Interventions: Biological: mRNA-1273
- Arm 10 (Experimental): 50 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age. N=15.
  Interventions: Biological: mRNA-1273
- Arm 11 (Experimental): 50 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 56-70 years of age. N=10.
  Interventions: Biological: mRNA-1273
- Arm 12 (Experimental): 50 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants 71 years of age or older. N=10.
  Interventions: Biological: mRNA-1273
- Arm 13 (Experimental): 10 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age. N=15.
  Interventions: Biological: mRNA-1273
- Arm 14 (Experimental): Optional third mRNA-1273 vaccination sub-study. 100 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle after Day 209 in participants from Arm 1,4,7,10, 11, and 12 from 18 years of age or older. N=70.
  Interventions: Biological: mRNA-1273
- Arm 15 (Experimental): Optional third mRNA-1273 vaccination sub-study. 100 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle no later than Day 394 in participants from Arm 2,3,5 and 8 from 18 years of age or older. N=50.
  Interventions: Biological: mRNA-1273
- Arm 2 (Experimental): 100 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age. N=15 (4 sentinel, 11 non-sentinel).
  Interventions: Biological: mRNA-1273
- Arm 3 (Experimental): 250 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age. N=15 (4 sentinel, 11 non-sentinel).
  Interventions: Biological: mRNA-1273
- Arm 4 (Experimental): 25 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 56-70 years of age. N=10.
  Interventions: Biological: mRNA-1273
- Arm 5 (Experimental): 100 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 56-70 years of age. N=10.
  Interventions: Biological: mRNA-1273
- Arm 6 (Experimental): 250 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 56-70 years of age. N=10.
  Interventions: Biological: mRNA-1273
- Arm 7 (Experimental): 25 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants 71 years of age or older. N=10.
  Interventions: Biological: mRNA-1273
- Arm 8 (Experimental): 100 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants 71 years of age or older. N=10.
  Interventions: Biological: mRNA-1273
- Arm 9 (Experimental): 250 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants 71 years of age or older. N=10.
  Interventions: Biological: mRNA-1273

INTERVENTIONS:
Biological: mRNA-1273 — Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.

SUMMARY:
This is a phase I, open-label, dose-ranging clinical trial in males and non-pregnant females, starting at 18 years of age, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of mRNA-1273 manufactured by ModernaTX, Inc. mRNA-1273 is a novel lipid nanoparticle (LNP)-encapsulated mRNA-based vaccine that encodes for a full-length, prefusion stabilized spike (S) protein of SARS-CoV-2. Enrollment will occur at up to 3 domestic clinical research sites. Up to one hundred and fifty-five subjects will be enrolled into one of thirteen cohorts (10 micrograms [mcg], 25 mcg, 50 mcg, 100 mcg, and 250 mcg). Subjects will receive an intramuscular (IM) injection (0.5 milliliters [mL]) of mRNA-1273 on Days 1 and 29 in the deltoid muscle and will be followed through 12 months post second vaccination (Day 394). Follow-up visits will occur 1, 2, and 4 weeks post each vaccination (Days 8, 15, 29, 36, 43, and 57), as well as 3, 6, and 12 months post second vaccination (Days 119, 209, and 394). The primary objective is to evaluate the safety and reactogenicity of a 2-dose vaccination schedule of mRNA-1273, given 28 days apart, across 5 dosages in healthy adults.

Optional Substudy:

This is an optional third mRNA-1273 vaccination substudy, in subjects 18 years of age and older, who received both the first and second mRNA-1273 vaccinations in the main study and meet all other substudy eligibility criteria. This optional third mRNA-1273 vaccination substudy is designed to assess safety, reactogenicity, and immunogenicity through 12 months post third vaccination (Day 731). Subjects who receive the third mRNA-1273 vaccination will exit the Schedule of Activities for the main study and will enter the Schedule of Activities for the optional substudy. Up to one hundred and twenty subject will be enrolled into two cohorts (consisting of participating subjects who received 2 doses of 25 or 50 mcg and participating subjects who received 2 doses of 100 and 250 mcg). Subjects will receive an IM injection (0.5 mL) at a dosage of 100 mcg/0.5 mL. The primary objective is to evaluate the safety and reactogenicity of a third mRNA-1273 vaccination, at a dosage of 100 mcg.

DETAILED DESCRIPTION:
This is a phase I, open-label, dose-ranging clinical trial in males and non-pregnant females, starting at 18 years of age, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of mRNA-1273 manufactured by ModernaTX, Inc. mRNA-1273 is a novel lipid nanoparticle (LNP)-encapsulated mRNA-based vaccine that encodes for a full-length, prefusion stabilized spike (S) protein of SARS-CoV-2. Enrollment will occur at up to 3 domestic clinical research sites. Up to one hundred and fifty-five subjects will be enrolled into one of thirteen cohorts (10 micrograms [mcg], 25 mcg, 50 mcg, 100 mcg, or 250 mcg). Subjects will receive an intramuscular (IM) injection (0.5 milliliters [mL]) of mRNA-1273 on Days 1 and 29 in the deltoid muscle and will be followed through 12 months post second vaccination (Day 394). Follow-up visits will occur 1, 2, and 4 weeks post each vaccination (Days 8, 15, 29, 36, 43, and 57), as well as 3, 6, and 12 months post second vaccination (Days 119, 209, and 394). The primary objective is to evaluate the safety and reactogenicity of a 2-dose vaccination schedule of mRNA-1273, given 28 days apart, across 5 dosages in healthy adults. The secondary objective is to evaluate the immunogenicity as measured by Immunoglobulin G (IgG) enzyme-linked immunosorbent assay (ELISA) to the SARS-CoV-2 S (spike) protein following a 2-dose vaccination schedule of mRNA-1273 at Day 57.

Optional Substudy:

This is an optional third mRNA-1273 vaccination substudy, in subjects 18 years of age and older, who received both the first and second mRNA-1273 vaccinations in the main study and meet all other substudy eligibility criteria. This optional third mRNA-1273 vaccination substudy is designed to assess safety, reactogenicity, and immunogenicity through 12 months post third vaccination (Day 731). Subjects who receive the third mRNA-1273 vaccination will exit the Schedule of Activities for the main study and will enter the Schedule of Activities for the optional substudy. Up to one hundred and twenty subject will be enrolled into two cohorts (consisting of participating subjects who received 2 doses of 25 or 50 mcg and participating subjects who received 2 doses of 100 and 250 mcg). Subjects will receive an IM injection (0.5 mL) at a dosage of 100 mcg/0.5 mL. The primary objective is to evaluate the safety and reactogenicity of a third mRNA-1273 vaccination, at a dosage of 100 mcg. The secondary objective is to evaluate the immunogenicity as measured by IgG ELISA to the SARS-CoV-2 S protein following a third mRNA-1273 vaccination, at a dosage of 100 mcg, at all timepoints after the third mRNA-1273 vaccination.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following criteria to be eligible to participate in this study:

1. Provides written informed consent prior to initiation of any study procedures.
2. Be able to understand and agrees to comply with planned study procedures and be available for all study visits.
3. Agrees to the collection of venous blood per protocol.
4. Male or non-pregnant female, >/= to 18 years of age at time of enrollment.
5. Body Mass Index (BMI) 18.0-35.0 kg/m^2, inclusive (< 56 years of age), at screening; BMI 18.0-30.0 kg/m^2, inclusive (>/= 56 years of age), at screening.
6. Women of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception.***, **** Note: These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).

   * Not of childbearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure(R) placement).

     * True abstinence is 100% of time no sexual intercourse (male's penis enters the female's vagina). (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

       * Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the subject's first vaccination, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products.

         * Must use at least one acceptable primary form of contraception for at least 30 days prior to the first vaccination and at least one acceptable primary form of contraception for 60 days after the last vaccination.
7. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to each vaccination.
8. Male subjects of childbearing potential*: use of condoms to ensure effective contraception with a female partner of childbearing potential from first vaccination until 60 days after the last vaccination.

   *Biological males who are post-pubertal and considered fertile until permanently sterile by bilateral orchiectomy or vasectomy.
9. Male subjects agree to refrain from sperm donation from the time of first vaccination until 60 days after the last vaccination.
10. In good health.* *As determined by medical history and physical examination to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of subjects. Chronic medical diagnoses/conditions should be stable for the last 60 days (no hospitalizations, emergency room (ER), or urgent care for condition or need for supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 60 days before enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the participating site principal investigator (PI) or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity, and do not indicate a worsening of medical diagnosis/condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided the change was not precipitated by deterioration in the chronic medical condition, and there is no anticipated additional risk to the subject or interference with the evaluation of responses to study vaccination.
11. Oral temperature is less than 100.0 degrees Fahrenheit (37.8 degrees Celsius).
12. Pulse no greater than 100 beats per minute.
13. Systolic blood pressure (BP) is 85 to 150 mm Hg, inclusive.
14. Clinical screening laboratory evaluations (white blood cell (WBC), hemoglobin (Hgb), platelets (PLTs), alanine transaminase (ALT), aspartate transaminase (AST), creatinine (Cr), alkaline phosphatase (ALP), total bilirubin (T. Bili), Lipase, prothrombin time (PT), and partial thromboplastin time (PTT)) are within acceptable normal reference ranges at the clinical laboratory being used.
15. Must agree to have samples stored for secondary research.
16. Agrees to adhere to Lifestyle Considerations throughout study duration.
17. Must agree to refrain from donating blood or plasma during the study (outside of this study).

Leukapheresis Inclusion Criteria:

A subject must meet all of the following criteria to be eligible for leukapheresis:

1. Written informed consent for leukapheresis is provided.
2. Weight >/= 110 pounds.
3. Screening laboratory evaluations are within acceptable ranges at the site where the leukapheresis procedure will be performed.
4. Negative urine or serum pregnancy test within 48 hours of the leukapheresis procedure for women of childbearing potential.
5. Adequate bilateral antecubital venous access.
6. No use of blood thinners, aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs) at least 5 days before the leukapheresis procedure.
7. Enrolled in cohorts 2, 3, 5, 10, or 11, and possibly cohort 6, if enrolled, and completed the two-dose vaccination series.

Optional Substudy Inclusion Criteria:

1. Enrolled in the main study and received both the first and second mRNA-1273 vaccinations.
2. Provides written informed consent for the third mRNA-1273 vaccination.
3. Agrees to the collection of venous blood per substudy.
4. Must agree to have samples stored for secondary research.
5. Women of childbearing potential have had a negative urine pregnancy test within 24 hours before the third mRNA-1273 vaccination.
6. Women of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception.***/****

   * Not of childbearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure® placement).

     * True abstinence is 100% of time no sexual intercourse (male's penis enters the female's vagina). (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

       * Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the subject's first vaccination, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products.

         ****Must use at least one acceptable primary form of contraception for at least 30 days prior to the third mRNA-1273 vaccination and for at least 30 days after the third mRNA-1273 vaccination.

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from participation in this study:

1. Positive pregnancy test either at screening or just prior to each vaccine administration.
2. Female subject who is breastfeeding or plans to breastfeed from the time of the first vaccination through 60 days after the last vaccination.
3. Has any medical disease or condition that, in the opinion of the participating site principal investigator (PI) or appropriate sub-investigator, precludes study participation.*

   *Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
4. Presence of self-reported or medically documented significant medical or psychiatric condition(s).*

   *Significant medical or psychiatric conditions include but are not limited to: Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma) requiring daily medications currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years. Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics.

   Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), history of myocarditis or pericarditis as an adult, myocardial infarction (MI) within past 6 months, coronary artery bypass surgery or stent placement, or uncontrolled cardiac arrhythmia.

   Neurological or neurodevelopmental conditions (e.g., history of migraines in the past 5 years, epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease).

   Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.

   An autoimmune disease, including hypothyroidism without a defined non-autoimmune cause, localized or history of psoriasis.

   An immunodeficiency of any cause. Chronic kidney disease, estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m^2.
5. Has an acute illness*, as determined by the participating site PI or appropriate sub-investigator, with or without fever [oral temperature >/= 38.0 degrees Celsius (100.4 degrees Fahrenheit)] within 72 hours prior to each vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
6. Has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) types 1 or 2 antibodies at screening.
7. Has participated in another investigational study involving any investigational product* within 60 days, or 5 half-lives, whichever is longer, before the first vaccine administration.

   *study drug, biologic or device
8. Currently enrolled in or plans to participate in another clinical trial with an investigational agent* that will be received during the study-reporting period.**

   *Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.

   **13 months after the first vaccination.
9. Has previously participated in an investigational study involving lipid nanoparticles (LNPs) (a component of the investigational vaccine assessed in this trial).
10. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to any previous licensed or unlicensed vaccines.
11. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness.*

    *Including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs during the preceding 6-month period prior to vaccine administration (Day 1). The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.
12. Anticipating the need for immunosuppressive treatment within the next 6 months.
13. Received immunoglobulins and/or any blood or blood products within the 4 months before the first vaccine administration or at any time during the study.
14. Has any blood dyscrasias or significant disorder of coagulation.
15. Has any chronic liver disease, including fatty liver.
16. Has a history of alcohol abuse or other recreational drug (excluding cannabis) use within 6 months before the first vaccine administration.
17. Has a positive test result for drugs of abuse at screening or before the first vaccine administration. If cannabis is the only detected drug, inclusion is permitted.
18. Has any abnormality or permanent body art (e.g., tattoo) that would interfere with the ability to observe local reactions at the injection site (deltoid region).
19. Received or plans to receive a licensed, live vaccine within 4 weeks before or after each vaccination.
20. Received or plans to receive a licensed, inactivated vaccine within 2 weeks before or after each vaccination.
21. Receipt of any other SARS-CoV-2 or other experimental coronavirus vaccine at any time prior to or during the study.
22. Close contact of anyone known to have SARS-CoV-2 infection within 30 days prior to vaccine administration.
23. History of COVID-19 diagnosis.
24. On current treatment with investigational agents for prophylaxis of COVID-19.
25. Current use of any prescription or over-the-counter medications within 7 days prior to vaccination, unless approved by the investigator or necessary to manage a chronic condition.
26. Plan to travel outside the United States (US) (continental US, Hawaii, and Alaska) from enrollment through 28 days after the last vaccination.
27. Reside in a nursing home or other skilled nursing facility or have a requirement for skilled nursing care.
28. Non-ambulatory.
29. For subjects >/= 56 years of age, history of chronic smoking within the prior year.
30. For subjects >/= 56 years of age, current smoking or vaping.
31. For subjects >/= 56 years of age, individuals currently working with high risk of exposure to SARS-CoV-2 (e.g., active health care workers with direct patient contact, emergency response personnel).

Optional Substudy Exclusion Criteria:

1. Anaphylaxis or other systemic hypersensitivity reaction following a mRNA-1273 or any other vaccination.
2. Immediate allergic reaction of any severity after mRNA-1273 or any of its components.*

   *Including polyethylene glycol (PEG)
3. Immediate allergic reaction of any severity to polysorbate.*

   *Due to potential cross-reactive hypersensitivity with the vaccine ingredient PEG
4. History of an SAE judged related to mRNA-1273 vaccine.
5. Female subject who is breastfeeding or plans to breastfeed from the time of the third mRNA-1273 vaccination through 30 days after the third mRNA-1273 vaccination.
6. Has an acute illness*, as determined by the participating site PI or appropriate sub-investigator, with or without fever [oral temperature >/=38.0°C (100.4°F)], within 72 hours prior to the third mRNA-1273 vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the substudy.
7. Has received any approved, authorized or investigational COVID-19 vaccine outside of this trial.
8. Any clinically significant medical condition that, in the opinion of the investigator, poses an additional risk to the subject from vaccination.
9. History of documented COVID-19 infection.
10. Has any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes substudy participation.
11. Received or plans to receive a licensed vaccine, other than a COVID-19 vaccine, within 2 weeks before or after the third mRNA-1273 vaccination.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Hope Clinic of Emory University, Decatur, Georgia
  - National Institutes of Health - Clinical Center - Vaccine Research Center Clinical Trials Program, Bethesda, Maryland
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington

REFERENCES:
- [Derived] Bangaru S, Jackson AM, Copps J, Fernandez-Quintero ML, Torres JL, Richey ST, Nogal B, Sewall LM, Torrents de la Pena A, Rehman A, Guebre-Xabier M, Girard B, Das R, Corbett-Helaire KS, Seder RA, Graham BS, Edwards DK, Patel N, Smith G, Ward AB. Structural serology of polyclonal antibody responses to mRNA-1273 and NVX-CoV2373 COVID-19 vaccines. Cell Rep. 2025 Jul 22;44(7):115986. doi: 10.1016/j.celrep.2025.115986. Epub 2025 Jul 8. PMID 40632654
- [Derived] Anderson E, Jackson L, Rouphael N, Widge A, Montefiori D, Doria-Rose N, Suthar M, Cohen K, O'Connell S, Makowski M, Makhene M, Buchanan W, Spearman P, Creech CB, O'Dell S, Schmidt S, Leav B, Bennett H, Pajon R, Posavad C, Hural J, Beigel J, Albert J, Abebe K, Eaton A, Rostad C, Rebolledo P, Kamidani S, Graciaa D, Coler R, McDermott A, Ledgerwood J, Mascola J, DeRosa S, Neuzil K, McElrath MJ, Roberts P. Safety and Immunogenicity of a Third Dose of SARS-CoV-2 mRNA Vaccine - An Interim Analysis. Res Sq [Preprint]. 2022 May 3:rs.3.rs-1222037. doi: 10.21203/rs.3.rs-1222037/v1. PMID 35547849
- [Derived] Jochum S, Kirste I, Hortsch S, Grunert VP, Legault H, Eichenlaub U, Kashlan B, Pajon R. Clinical Utility of Elecsys Anti-SARS-CoV-2 S Assay in COVID-19 Vaccination: An Exploratory Analysis of the mRNA-1273 Phase 1 Trial. Front Immunol. 2022 Jan 19;12:798117. doi: 10.3389/fimmu.2021.798117. eCollection 2021. PMID 35126362
- [Derived] Garrett ME, Galloway JG, Wolf C, Logue JK, Franko N, Chu HY, Matsen FA 4th, Overbaugh JM. Comprehensive characterization of the antibody responses to SARS-CoV-2 Spike protein finds additional vaccine-induced epitopes beyond those for mild infection. Elife. 2022 Jan 24;11:e73490. doi: 10.7554/eLife.73490. PMID 35072628
- [Derived] Jochum S, Kirste I, Hortsch S, Grunert VP, Legault H, Eichenlaub U, Kashlan B, Pajon R. Clinical utility of Elecsys Anti-SARS-CoV-2 S assay in COVID-19 vaccination: An exploratory analysis of the mRNA-1273 phase 1 trial. medRxiv [Preprint]. 2021 Oct 19:2021.10.04.21264521. doi: 10.1101/2021.10.04.21264521. PMID 34642699
- [Derived] Mendes BB, Sousa DP, Conniot J, Conde J. Nanomedicine-based strategies to target and modulate the tumor microenvironment. Trends Cancer. 2021 Sep;7(9):847-862. doi: 10.1016/j.trecan.2021.05.001. Epub 2021 Jun 3. PMID 34090865
- [Derived] Anderson EJ, Rouphael NG, Widge AT, Jackson LA, Roberts PC, Makhene M, Chappell JD, Denison MR, Stevens LJ, Pruijssers AJ, McDermott AB, Flach B, Lin BC, Doria-Rose NA, O'Dell S, Schmidt SD, Corbett KS, Swanson PA 2nd, Padilla M, Neuzil KM, Bennett H, Leav B, Makowski M, Albert J, Cross K, Edara VV, Floyd K, Suthar MS, Martinez DR, Baric R, Buchanan W, Luke CJ, Phadke VK, Rostad CA, Ledgerwood JE, Graham BS, Beigel JH; mRNA-1273 Study Group. Safety and Immunogenicity of SARS-CoV-2 mRNA-1273 Vaccine in Older Adults. N Engl J Med. 2020 Dec 17;383(25):2427-2438. doi: 10.1056/NEJMoa2028436. Epub 2020 Sep 29. PMID 32991794
- [Derived] Jackson LA, Anderson EJ, Rouphael NG, Roberts PC, Makhene M, Coler RN, McCullough MP, Chappell JD, Denison MR, Stevens LJ, Pruijssers AJ, McDermott A, Flach B, Doria-Rose NA, Corbett KS, Morabito KM, O'Dell S, Schmidt SD, Swanson PA 2nd, Padilla M, Mascola JR, Neuzil KM, Bennett H, Sun W, Peters E, Makowski M, Albert J, Cross K, Buchanan W, Pikaart-Tautges R, Ledgerwood JE, Graham BS, Beigel JH; mRNA-1273 Study Group. An mRNA Vaccine against SARS-CoV-2 - Preliminary Report. N Engl J Med. 2020 Nov 12;383(20):1920-1931. doi: 10.1056/NEJMoa2022483. Epub 2020 Jul 14. PMID 32663912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited for this study include males and non-pregnant females of 18 or more years of age, who were in good health and met all eligibility criteria. Participants were recruited from the community surrounding the clinical sites. Enrollment occurred between 16MAR2020 and 17JUNE2020.
Groups:
- 10 mcg of mRNA-1273: 18-55 Years: 10 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 25 mcg of mRNA-1273: 18-55 Years: 25 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 50 mcg of mRNA-1273:18-55 Years: 50 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 100 mcg of mRNA-1273: 18-55 Years: 100 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 250 mcg of mRNA-1273: 18-55 Years: 250 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 18-55 years of age.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 25 mcg of mRNA-1273: 56-70 Years: 25 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 56-70 years of age.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 50 mcg of mRNA-1273: 56-70 Years: 50 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 56-70 years of age.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 100 mcg of mRNA-1273: 56-70 Years: 100 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 56-70 years of age.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 250 mcg of mRNA-1273: 56-70 Years: 250 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants from 56-70 years of age.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 25 mcg of mRNA-1273: 71+ Years: 25 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants 71 years of age or older.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 50 mcg of mRNA-1273: 71+ Years: 50 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants 71 years of age or older.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 100 mcg of mRNA-1273: 71+ Years: 100 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants 71 years of age or older.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
- 250 mcg of mRNA-1273: 71+ Years: 250 mcg of mRNA-1273 administered through 0.5 mL intramuscular injection in the deltoid muscle on Days 1 and 29 in participants 71 years of age or older.
  mRNA-1273: Lipid nanoparticle (LNP) dispersion containing an mRNA that encodes for the prefusion stabilized spike protein 2019-nCoV. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, DSPC, and PEG2000 DMG.
Period: Overall Study
Arm/Group | 10 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 250 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years | 250 mcg of mRNA-1273: 71+ Years
Started | 0 | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 0 | 10 | 10 | 10 | 0
Completed | 0 | 15 | 7 | 2 | 3 | 10 | 10 | 2 | 0 | 10 | 10 | 3 | 0
Not Completed | 0 | 0 | 8 | 13 | 12 | 0 | 0 | 8 | 0 | 0 | 0 | 7 | 0
Not completed — Enrolled in separate trial | 0 | 0 | 8 | 13 | 12 | 0 | 0 | 8 | 0 | 0 | 0 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- 25 mcg of mRNA-1273: 18-55 Years: 25 mcg of mRNA-1273 administered on Days 1 and 29 in participants from 18-55 years of age.
- 50 mcg of mRNA-1273:18-55 Years: 50 mcg of mRNA-1273 administered on Days 1 and 29 in participants from 18-55 years of age.
- 100 mcg of mRNA-1273: 18-55 Years: 100 mcg of mRNA-1273 administered on Days 1 and 29 in participants from 18-55 years of age.
- 250 mcg of mRNA-1273: 18-55 Years: 250 mcg of mRNA-1273 administered on Days 1 and 29 in participants from 18-55 years of age.
- 25 mcg of mRNA-1273: 56-70 Years: 25 mcg of mRNA-1273 administered on Days 1 and 29 in participants from 56-70 years of age.
- 50 mcg of mRNA-1273: 56-70 Years: 50 mcg of mRNA-1273 administered on Days 1 and 29 in participants from 56-70 years of age.
- 100 mcg of mRNA-1273: 56-70 Years: 100 mcg of mRNA-1273 administered on Days 1 and 29 in participants from 56-70 years of age.
- 25 mcg of mRNA-1273: 71+ Years: 25 mcg of mRNA-1273 administered on Days 1 and 29 in participants 71 years of age or older.
- 50 mcg of mRNA-1273: 71+ Years: 50 mcg of mRNA-1273 administered on Days 1 and 29 in participants 71 years of age or older.
- 100 mcg of mRNA-1273: 71+ Years: 100 mcg of mRNA-1273 administered on Days 1 and 29 in participants 71 years of age or older.
- Total: Total of all reporting groups
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (8.0) | 36.5 (9.9) | 30.8 (8.9) | 30.4 (8.0) | 65.4 (4.6) | 61.6 (3.7) | 63.3 (4.2) | 72.3 (1.3) | 74.7 (3.5) | 72.2 (1.2) | 51.3 (19.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 8 | 9 | 7 | 5 | 5 | 2 | 4 | 7 | 59
  Male | 9 | 9 | 7 | 6 | 3 | 5 | 5 | 8 | 6 | 3 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 9
  Not Hispanic or Latino | 14 | 14 | 12 | 13 | 10 | 10 | 10 | 9 | 9 | 10 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  White | 15 | 13 | 11 | 14 | 10 | 7 | 10 | 9 | 10 | 10 | 109
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10 | 120

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Any Medically-attended Adverse Events (MAAEs)
Description: Number of participants that experienced any MAAEs from Day 1 to Day 394.
Time Frame: Day 1 to Day 394
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
Participants | 7 | 6 | 5 | 7 | 2 | 6 | 2 | 5 | 4 | 8

2. Primary Outcome: Frequency of Any New-onset Chronic Medical Conditions (NOCMCs)
Description: Number of participants that experienced any NOCMCs from Day 1 to Day 394.
Time Frame: Day 1 to Day 394
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
Participants | 0 | 0 | 2 | 2 | 1 | 3 | 0 | 0 | 1 | 1

3. Primary Outcome: Frequency of Any Serious Adverse Events (SAEs)
Description: The number of participants that experience any SAEs from Day 1 to Day 394. An AE or suspected adverse reaction is considered serious if, in the view of either the participating site PI or appropriate sub-investigator or the sponsor, it results in: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 to Day 394
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Frequency of Solicited Reactogenicity Adverse Events (AEs)
Description: The number of participants that experienced at least one solicited (local and systemic) AE through 7 days post vaccination. Systemic events include: fatigue, headache, myalgia, arthralgia, nausea, chills and fever. Local events include: pain at injection site, erythema, and induration.
Time Frame: Through 7 days post-vaccination
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Number; unit: participants
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
participants
  Local Events | 11 | 14 | 15 | 15 | 8 | 9 | 9 | 8 | 7 | 10
  Systemic Events | 8 | 13 | 15 | 15 | 8 | 6 | 8 | 5 | 6 | 7

5. Primary Outcome: Frequency of Any Unsolicited Adverse Events (AEs) by Relationship to Study Product and Severity
Description: Number of events of any unsolicited AE through 28 days post vaccination by relationship to study product and severity, experienced by participants in the Safety Analysis population . Unsolicited AEs were events that were spontaneously reported by the subject, or revealed by observation, physical examination or other diagnostic procedures.
Time Frame: Through 28 days post-vaccination
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Number; unit: events
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
events
  Not Related : Mild | 28 | 22 | 15 | 16 | 9 | 6 | 5 | 18 | 8 | 26
  Not Related : Moderate | 3 | 7 | 6 | 14 | 7 | 4 | 7 | 5 | 6 | 4
  Not Related : Severe | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
  Related : Mild | 4 | 5 | 10 | 11 | 2 | 0 | 1 | 12 | 2 | 3
  Related : Moderate | 1 | 1 | 3 | 7 | 2 | 1 | 0 | 0 | 0 | 0
  Related : Severe | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Grade of Any Unsolicited Adverse Events (AEs)
Description: Number of any unsolicited AEs through 28 days post vaccination by severity
Time Frame: Through 28 days post-vaccination
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Number; unit: events
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
events
  Mild | 32 | 27 | 25 | 27 | 11 | 6 | 6 | 30 | 10 | 29
  Moderate | 4 | 8 | 9 | 21 | 9 | 5 | 7 | 5 | 6 | 4
  Severe | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 0

7. Primary Outcome: Grade of Solicited Reactogenicity Adverse Events (AEs)
Description: Number of participants who experienced any solicited (local and systemic) AEs through 7 days post vaccination by grade. Systemic events include: fatigue, headache, myalgia, arthralgia, nausea, chills and fever. Local events include: pain at injection site, erythema, and induration.
Time Frame: Through 7 days post vaccination
Population: The Safety Analysis population for the main study includes all participants who received one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
Participants
  Dose 1: None | 5 | 0 | 1 | 0 | 3 | 4 | 1 | 1 | 2 | 2
  Dose 1: Mild | 8 | 10 | 10 | 9 | 5 | 4 | 9 | 9 | 7 | 8
  Dose 1: Moderate | 2 | 5 | 3 | 5 | 2 | 2 | 0 | 0 | 1 | 0
  Dose 1: Severe | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: number analyzed (Participants) | 13 | 15 | 15 | 14 | 10 | 10 | 9 | 10 | 10 | 10
  Dose 2: None | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 0
  Dose 2: Mild | 7 | 7 | 3 | 2 | 7 | 7 | 2 | 7 | 6 | 6
  Dose 2: Moderate | 3 | 7 | 11 | 8 | 2 | 0 | 6 | 2 | 1 | 3
  Dose 2: Severe | 0 | 1 | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 1

8. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in IgG Titer From Baseline Against RBD
Description: Geometric mean fold rise (GMFR) in IgG ELISA titer from baseline against RBD. Fold-rise is calculated by dividing post-vaccination results by the baseline value.
Time Frame: Day 1 to Day 394
Population: The modified intent-to-treat (mITT) population includes all participants who received one dose of vaccine and contributed both pre- and at least one post-vaccination venous blood samples for immunogenicity testing for which valid results were reported.
Measure: Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
Fold Rise
  Day 15 | 118.232 [60.888 to 229.579] | 46.423 [24.502 to 87.956] | 205.148 [105.848 to 397.603] | 151.985 [74.288 to 310.944] | 14.358 [2.731 to 75.481] | 24.082 [12.174 to 47.639] | 138.867 [47.290 to 407.785] | 42.034 [14.335 to 123.258] | 11.013 [2.664 to 45.534] | 51.027 [17.037 to 152.833]
  Day 29: number analyzed (Participants) | 15 | 15 | 15 | 14 | 10 | 10 | 10 | 10 | 10 | 10
  Day 29 | 326.688 [194.477 to 548.780] | 113.292 [51.591 to 248.785] | 561.479 [264.946 to 1189.896] | 222.148 [107.069 to 460.915] | 23.779 [5.816 to 97.219] | 38.967 [19.884 to 76.363] | 204.880 [54.672 to 767.772] | 137.911 [37.221 to 510.994] | 42.530 [11.332 to 159.622] | 112.047 [39.432 to 318.385]
  Day 36 | 2621.803 [1355.412 to 5071.410] | 1122.191 [669.513 to 1880.939] | 3007.923 [1610.324 to 5618.496] | 1086.092 [554.012 to 2129.187] | 975.663 [330.190 to 2882.945] | 303.529 [136.134 to 676.756] | 4418.756 [1818.818 to 10735.216] | 1443.444 [386.453 to 5391.417] | 407.474 [109.921 to 1510.502] | 1414.165 [487.854 to 4099.307]
  Day 43: number analyzed (Participants) | 15 | 14 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 43 | 2734.849 [1338.670 to 5587.186] | 1073.107 [726.428 to 1585.232] | 3527.768 [1637.665 to 7599.321] | 941.022 [437.492 to 2024.092] | 989.692 [411.218 to 2381.921] | 701.940 [272.166 to 1810.366] | 3071.850 [1480.126 to 6375.312] | 2653.994 [759.931 to 9268.852] | 657.204 [173.073 to 2495.569] | 1380.702 [475.775 to 4006.810]
  Day 57: number analyzed (Participants) | 15 | 15 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 57 | 2427.728 [1238.979 to 4757.030] | 877.135 [557.842 to 1379.184] | 2343.458 [963.830 to 5697.890] | 839.589 [364.917 to 1931.696] | 383.266 [156.920 to 936.101] | 578.229 [249.207 to 1341.649] | 1611.388 [367.006 to 7075.003] | 1962.908 [480.835 to 8013.154] | 626.325 [180.467 to 2173.714] | 901.571 [270.733 to 3002.336]
  Day 119 | 1707.917 [793.649 to 3675.400] | 195.764 [117.352 to 326.571] | 1416.229 [684.896 to 2928.480] | 346.524 [164.750 to 728.856] | 223.100 [82.918 to 600.274] | 154.917 [61.416 to 390.765] | 463.340 [141.681 to 1515.262] | 593.198 [150.885 to 2332.137] | 187.845 [59.459 to 593.450] | 313.979 [88.410 to 1115.058]
  Day 209: number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 9 | 10 | 10 | 10 | 9
  Day 209 | 368.468 [187.618 to 723.644] | 40.957 [23.071 to 72.712] | 556.673 [290.404 to 1067.082] | 91.215 [44.456 to 187.154] | 100.000 [33.500 to 298.509] | 285.832 [140.919 to 579.766] | 181.844 [55.959 to 590.924] | 201.187 [52.192 to 775.526] | 475.445 [153.101 to 1476.465] | 91.951 [27.684 to 305.406]
  Day 394: number analyzed (Participants) | 15 | 12 | 14 | 15 | 7 | 10 | 10 | 10 | 10 | 10
  Day 394 | 727.556 [399.079 to 1326.400] | 190.546 [51.219 to 708.876] | 441.135 [110.864 to 1755.303] | 61.113 [31.403 to 118.932] | 79.878 [11.702 to 545.251] | 114.078 [31.552 to 412.448] | 183.781 [39.490 to 855.284] | 285.957 [31.077 to 2631.214] | 451.648 [113.720 to 1793.750] | 110.892 [26.367 to 466.386]

9. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in IgG Titer From Baseline Against S-2
Description: Geometric mean fold rise (GMFR) in IgG titer from baseline against S-2P (Wa-1). Fold-rise is calculated by dividing post-vaccination results by the baseline value.
Time Frame: Day 1 to Day 394
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
Fold Rise
  Day 15 | 278.826 [120.686 to 644.185] | 190.575 [92.860 to 391.117] | 656.649 [327.031 to 1318.492] | 915.658 [418.876 to 2001.617] | 55.693 [9.591 to 323.405] | 78.037 [39.479 to 154.251] | 84.723 [33.765 to 212.586] | 133.721 [54.358 to 328.953] | 20.706 [6.404 to 66.946] | 109.977 [31.717 to 381.332]
  Day 29: number analyzed (Participants) | 15 | 15 | 15 | 14 | 10 | 10 | 10 | 10 | 10 | 10
  Day 29 | 347.590 [170.815 to 707.305] | 334.452 [129.835 to 861.536] | 830.870 [379.340 to 1819.858] | 1259.340 [532.930 to 2975.879] | 93.735 [16.091 to 546.028] | 79.671 [35.902 to 176.798] | 176.685 [61.056 to 511.295] | 522.637 [177.450 to 1539.307] | 49.900 [15.513 to 160.514] | 213.206 [102.237 to 444.622]
  Day 36 | 2497.277 [1278.098 to 4879.431] | 2450.191 [828.251 to 7248.329] | 5943.834 [2823.630 to 12511.967] | 6601.865 [2948.586 to 14781.533] | 1662.647 [446.013 to 6198.010] | 358.509 [157.061 to 818.338] | 4779.693 [543.021 to 42071.027] | 4145.720 [1610.338 to 10672.911] | 297.577 [97.440 to 908.791] | 2765.031 [796.460 to 9599.223]
  Day 43: number analyzed (Participants) | 15 | 14 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 43 | 2425.121 [1306.938 to 4499.992] | 2512.713 [1008.639 to 6259.647] | 6380.536 [2845.471 to 14307.382] | 5007.258 [2114.555 to 11857.170] | 2523.481 [856.050 to 7438.764] | 744.903 [390.710 to 1420.187] | 1548.460 [315.724 to 7594.384] | 2737.159 [913.784 to 8198.917] | 774.819 [213.610 to 2810.468] | 8483.987 [2252.065 to 31960.904]
  Day 57: number analyzed (Participants) | 15 | 15 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 57 | 1976.059 [982.475 to 3974.462] | 1588.791 [666.141 to 3789.374] | 6157.842 [3199.803 to 11850.426] | 6479.378 [2562.589 to 16382.782] | 1715.932 [428.208 to 6876.149] | 559.114 [319.663 to 977.930] | 1393.157 [251.085 to 7729.989] | 10169.509 [3720.365 to 27798.057] | 483.727 [164.214 to 1424.920] | 3815.048 [1262.647 to 11527.051]
  Day 119 | 1964.265 [1092.299 to 3532.306] | 511.132 [162.699 to 1605.762] | 3148.715 [1628.418 to 6088.368] | 3190.558 [1258.565 to 8088.311] | 457.931 [131.073 to 1599.876] | 134.834 [68.773 to 264.353] | 385.745 [95.962 to 1550.604] | 682.182 [271.806 to 1712.148] | 184.289 [51.001 to 665.918] | 204.739 [102.957 to 407.139]
  Day 209: number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 9 | 10 | 10 | 10 | 9
  Day 209 | 532.926 [259.219 to 1095.636] | 349.194 [133.310 to 914.681] | 639.244 [330.763 to 1235.426] | 391.021 [164.947 to 926.949] | 149.796 [41.609 to 539.277] | 127.513 [64.754 to 251.097] | 131.644 [31.225 to 554.998] | 374.024 [148.317 to 943.210] | 193.464 [64.217 to 582.841] | 114.639 [42.789 to 307.141]
  Day 394: number analyzed (Participants) | 15 | 12 | 14 | 15 | 7 | 10 | 10 | 10 | 10 | 10
  Day 394 | 467.448 [196.093 to 1114.309] | 426.170 [157.075 to 1156.273] | 1079.124 [360.017 to 3234.598] | 650.429 [219.338 to 1928.793] | 217.986 [25.301 to 1878.122] | 214.487 [53.375 to 861.917] | 258.048 [80.107 to 831.244] | 824.518 [106.753 to 6368.232] | 824.138 [160.041 to 4243.928] | 50.304 [22.538 to 112.273]

10. Secondary Outcome: Geometric Mean Titer (GMT) of Antibody Against RBD
Description: Geometric mean titer (GMT) of antibody against RBD
Time Frame: Day 1 to Day 394
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Titer
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
Titer
  Day 1 | 55.539 [44.340 to 69.567] | 588.031 [411.408 to 840.480] | 166.061 [81.760 to 337.282] | 575.528 [349.084 to 948.863] | 203.610 [113.648 to 364.785] | 348.980 [165.342 to 736.573] | 223.049 [64.175 to 775.238] | 111.224 [45.771 to 270.276] | 193.821 [92.028 to 408.205] | 503.037 [174.025 to 1454.084]
  Day 15 | 6566.491 [3650.209 to 11812.694] | 27298.157 [15906.715 to 46847.473] | 34066.956 [21684.705 to 53519.636] | 87471.519 [51857.424 to 147544.285] | 2923.479 [576.391 to 14828.010] | 8404.270 [5860.592 to 12051.983] | 30974.193 [15895.840 to 60355.452] | 4675.198 [2235.438 to 9777.713] | 2134.519 [513.626 to 8870.598] | 25668.471 [12391.568 to 53170.866]
  Day 29: number analyzed (Participants) | 15 | 15 | 15 | 14 | 10 | 10 | 10 | 10 | 10 | 10
  Day 29 | 18144.012 [11088.170 to 29689.766] | 66619.290 [35965.306 to 123400.305] | 93239.514 [59894.633 to 145148.347] | 120088.107 [71026.274 to 203039.702] | 4841.724 [1531.597 to 15305.782] | 13598.782 [7948.752 to 23264.892] | 45698.295 [26323.563 to 79333.264] | 15339.104 [7087.422 to 33197.985] | 8243.279 [2486.083 to 27332.811] | 56363.766 [35061.830 to 90607.766]
  Day 36 | 145612.950 [77796.145 to 272547.326] | 659882.584 [466389.271 to 933651.463] | 499497.517 [400839.447 to 622438.163] | 625076.733 [437605.395 to 892861.300] | 198655.229 [98717.264 to 399766.951] | 105925.373 [50971.843 to 220125.148] | 985598.423 [284610.485 to 3413100.720] | 160546.189 [82581.200 to 312117.997] | 78976.885 [25690.683 to 242786.399] | 711377.295 [368425.491 to 1373568.519]
  Day 43: number analyzed (Participants) | 15 | 14 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 43 | 151891.452 [74930.671 to 307898.124] | 572701.831 [398614.411 to 822818.689] | 558929.643 [462950.139 to 674807.758] | 541585.049 [347184.872 to 844836.250] | 201511.576 [115921.617 to 350296.315] | 244962.722 [154477.301 to 388450.181] | 685172.620 [222613.551 to 2108863.173] | 295188.885 [167304.797 to 520824.741] | 127379.635 [44079.970 to 368093.979] | 694544.378 [465009.324 to 1037381.118]
  Day 57: number analyzed (Participants) | 15 | 15 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 57 | 134834.181 [70747.115 to 256975.230] | 515782.576 [328490.907 to 809860.058] | 371290.883 [266713.944 to 516871.813] | 483207.129 [303572.459 to 769138.051] | 78036.898 [42855.978 to 142098.203] | 201790.167 [135955.705 to 299503.957] | 359418.146 [128908.940 to 1002113.613] | 218323.256 [106760.447 to 446467.258] | 121394.777 [43523.048 to 338595.123] | 453523.713 [255612.038 to 804671.643]
  Day 119 | 94856.406 [44231.293 to 203424.707] | 115115.375 [75506.457 to 175502.205] | 235179.791 [177210.044 to 312112.863] | 199434.367 [127702.777 to 311458.121] | 45425.530 [23050.545 to 89519.739] | 54062.982 [36881.823 to 79247.873] | 103347.506 [38416.686 to 278022.601] | 65978.130 [33230.207 to 130998.691] | 36408.266 [15287.605 to 86708.273] | 157942.861 [94323.027 to 264473.564]
  Day 209: number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 9 | 10 | 10 | 10 | 9
  Day 209 | 20464.446 [10276.948 to 40750.773] | 24084.261 [14896.240 to 38939.467] | 92441.432 [57141.666 to 149547.939] | 52496.861 [34936.109 to 78884.582] | 20361.042 [9275.521 to 44695.280] | 123784.614 [69755.695 to 219661.357] | 40560.192 [13771.075 to 119462.654] | 22376.904 [11234.479 to 44570.454] | 92150.989 [35818.319 to 237079.938] | 49367.876 [25170.231 to 96828.163]
  Day 394: number analyzed (Participants) | 15 | 12 | 14 | 15 | 7 | 10 | 10 | 10 | 10 | 10
  Day 394 | 40407.936 [23427.721 to 69695.268] | 90573.260 [27756.903 to 295548.658] | 70794.578 [30435.905 to 164669.732] | 35172.238 [20744.761 to 59633.674] | 12844.414 [3233.887 to 51015.689] | 39810.717 [17869.264 to 88693.813] | 40992.084 [14189.286 to 118423.929] | 31805.337 [4545.268 to 222556.593] | 87538.681 [35329.764 to 216899.856] | 55782.760 [13635.712 to 228203.428]

11. Secondary Outcome: Geometric Mean Titer (GMT) of Antibody Against S-2P
Description: Geometric mean titer (GMT) of antibody against S-2P (Wa-1)
Time Frame: Day 1 to Day 394
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Titer
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
Titer
  Day 1 | 115.700 [71.727 to 186.630] | 353.726 [132.208 to 946.402] | 131.442 [64.973 to 265.910] | 178.484 [81.254 to 392.061] | 188.712 [76.456 to 465.788] | 563.378 [315.579 to 1005.753] | 655.541 [270.066 to 1591.222] | 110.943 [55.418 to 222.100] | 324.564 [103.755 to 1015.294] | 953.674 [493.489 to 1842.990]
  Day 15 | 32260.171 [18721.778 to 55588.665] | 67411.398 [32440.518 to 140080.890] | 86311.103 [56413.130 to 132054.478] | 163430.584 [102144.589 to 261487.722] | 10509.934 [2841.259 to 38876.682] | 43964.284 [20823.983 to 92818.854] | 55539.249 [40604.778 to 75966.629] | 14835.425 [6923.655 to 31788.101] | 6720.475 [1734.084 to 26045.329] | 104881.768 [22438.517 to 490236.733]
  Day 29: number analyzed (Participants) | 15 | 15 | 15 | 14 | 10 | 10 | 10 | 10 | 10 | 10
  Day 29 | 40216.104 [29088.696 to 55600.122] | 118304.156 [71951.240 to 194518.861] | 109211.071 [79048.399 to 150882.981] | 213515.089 [128810.327 to 353921.103] | 17688.866 [5303.052 to 59003.006] | 44884.873 [23416.011 to 86037.364] | 115824.384 [73271.749 to 183089.502] | 57982.909 [31454.265 to 106885.911] | 16195.710 [5218.359 to 50265.040] | 203329.316 [97384.457 to 424531.922]
  Day 36 | 288934.898 [166075.942 to 502681.932] | 866695.749 [641509.478 to 1170928.175] | 781267.935 [606074.064 to 1007103.952] | 1178329.272 [889033.807 to 1561762.739] | 313761.751 [160505.758 to 613351.431] | 201976.108 [99730.675 to 409045.145] | 3133285.724 [570561.057 to 17206711.371] | 459938.749 [272869.372 to 775256.128] | 96582.846 [39661.176 to 235198.426] | 2636938.493 [1072568.674 to 6482983.127]
  Day 43: number analyzed (Participants) | 15 | 14 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 43 | 280586.432 [167983.735 to 468668.862] | 734030.804 [588265.571 to 915914.933] | 811094.448 [656186.213 to 1002572.427] | 893716.961 [661380.499 to 1207670.935] | 476211.633 [264023.482 to 858929.354] | 419662.342 [303128.058 to 580996.964] | 1015079.367 [408139.653 to 2524592.041] | 303668.679 [167756.794 to 549692.591] | 251478.001 [119947.760 to 527239.400] | 8090958.992 [2546021.264 to 25712125.163]
  Day 57: number analyzed (Participants) | 15 | 15 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 57 | 228630.062 [134203.687 to 389495.298] | 561996.141 [407302.734 to 775442.039] | 782785.653 [619387.634 to 989289.008] | 1156467.236 [859119.097 to 1556729.996] | 323817.265 [182136.112 to 575710.221] | 314992.345 [217858.591 to 455433.854] | 913271.700 [287340.911 to 2902702.559] | 1128236.122 [635868.259 to 2001856.089] | 157000.126 [81997.547 to 300607.036] | 3638312.512 [1315790.941 to 10060350.416]
  Day 119 | 227265.406 [137995.234 to 374285.134] | 180800.655 [109897.259 to 297449.430] | 413872.592 [322840.850 to 530572.641] | 569464.514 [422292.607 to 767926.854] | 86417.162 [51215.401 to 145814.068] | 75962.631 [52415.295 to 110088.503] | 252871.567 [96427.352 to 663131.657] | 75683.290 [53033.587 to 108006.278] | 59813.608 [32284.811 to 110815.815] | 195254.027 [117658.578 to 324023.422]
  Day 209: number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 9 | 10 | 10 | 10 | 9
  Day 209 | 61659.500 [34984.758 to 108672.866] | 123518.877 [75876.495 to 201075.616] | 84023.351 [60469.283 to 116752.229] | 69791.093 [52610.682 to 92581.896] | 28268.320 [14750.596 to 54173.939] | 74683.080 [55359.100 to 100752.405] | 86297.855 [34927.116 to 213224.580] | 41495.404 [31129.203 to 55313.610] | 62791.376 [32873.371 to 119937.712] | 112287.997 [57588.133 to 218944.311]
  Day 394: number analyzed (Participants) | 15 | 12 | 14 | 15 | 7 | 10 | 10 | 10 | 10 | 10
  Day 394 | 54083.734 [29885.281 to 97875.950] | 115722.196 [48958.299 to 273531.291] | 151979.746 [65657.023 to 351795.467] | 116091.387 [57500.772 to 234383.115] | 44800.794 [6793.925 to 295427.350] | 120837.018 [43121.651 to 338613.777] | 169160.905 [75032.538 to 381373.369] | 91474.491 [17505.769 to 477990.007] | 267485.349 [100394.424 to 712673.167] | 47973.345 [24336.780 to 94566.406]

12. Secondary Outcome: Percentage of Participants Who Seroconverted Against RBD
Description: Percentage of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against RBD
Time Frame: Day 1 to Day 394
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
percentage of participants
  Day 15 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 60 [26.2 to 87.8] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 90 [55.5 to 99.7] | 60 [26.2 to 87.8] | 90 [55.5 to 99.7]
  Day 29: number analyzed (Participants) | 15 | 15 | 15 | 14 | 10 | 10 | 10 | 10 | 10 | 10
  Day 29 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [76.8 to 100.0] | 80 [44.4 to 97.5] | 100 [69.2 to 100.0] | 90 [55.5 to 99.7] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]
  Day 36 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]
  Day 43: number analyzed (Participants) | 15 | 14 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 43 | 100 [78.2 to 100.0] | 100 [76.8 to 100.0] | 100 [76.8 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]
  Day 57: number analyzed (Participants) | 15 | 15 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 57 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [76.8 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]
  Day 119 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]
  Day 209: number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 9 | 10 | 10 | 10 | 9
  Day 209 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [66.4 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [66.4 to 100.0]
  Day 394: number analyzed (Participants) | 15 | 12 | 14 | 15 | 7 | 10 | 10 | 10 | 10 | 10
  Day 394 | 100 [78.2 to 100.0] | 100 [73.5 to 100.0] | 100 [76.8 to 100.0] | 100 [78.2 to 100.0] | 100 [59.0 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 90 [55.5 to 99.7] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]

13. Secondary Outcome: Percentage of Participants Who Seroconverted Against S-2P
Description: Percentage of participants who seroconverted defined as a 4-fold change in antibody titer from baseline against S-2P (Wa-1)
Time Frame: Day 1 to Day 394
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 10 | 10 | 10 | 10 | 10
percentage of participants
  Day 15 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 90 [55.5 to 99.7] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 90 [55.5 to 99.7] | 100 [69.2 to 100.0]
  Day 29: number analyzed (Participants) | 15 | 15 | 15 | 14 | 10 | 10 | 10 | 10 | 10 | 10
  Day 29 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [76.8 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 90 [55.5 to 99.7] | 100 [69.2 to 100.0]
  Day 36 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]
  Day 43: number analyzed (Participants) | 15 | 14 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 43 | 100 [78.2 to 100.0] | 100 [76.8 to 100.0] | 100 [76.8 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]
  Day 57: number analyzed (Participants) | 15 | 15 | 14 | 15 | 10 | 10 | 10 | 10 | 10 | 10
  Day 57 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [76.8 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]
  Day 119 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]
  Day 209: number analyzed (Participants) | 15 | 15 | 15 | 15 | 10 | 9 | 10 | 10 | 10 | 9
  Day 209 | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [78.2 to 100.0] | 100 [69.2 to 100.0] | 100 [66.4 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [66.4 to 100.0]
  Day 394: number analyzed (Participants) | 15 | 12 | 14 | 15 | 7 | 10 | 10 | 10 | 10 | 10
  Day 394 | 100 [78.2 to 100.0] | 100 [73.5 to 100.0] | 100 [76.8 to 100.0] | 100 [78.2 to 100.0] | 100 [59.0 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0] | 100 [69.2 to 100.0]

ADVERSE EVENTS:
Time Frame: Solicited (local and systemic) AEs were collected Day 1 through 7 days post vaccination (Days 1-8 and Days 29-36); Unsolicited AEs were collected from Day 1 through 28 days post second vaccination (Days 1-57); SAEs, MAAEs, and NOCMCs were collected from Day 1 through the end of the study (Days 1-394).
Description: Systemic AEs include fatigue, headache, myalgia, arthralgia, nausea, chills and fever. Local events include: pain at injection site, erythema, and induration. Unsolicited AEs were all AEs spontaneously reported by the subject and/or in response to an open question from study staff or revealed by observation, physical examination or other diagnostic procedures.
Arm/Group | 25 mcg of mRNA-1273: 18-55 Years | 50 mcg of mRNA-1273:18-55 Years | 100 mcg of mRNA-1273: 18-55 Years | 250 mcg of mRNA-1273: 18-55 Years | 25 mcg of mRNA-1273: 56-70 Years | 50 mcg of mRNA-1273: 56-70 Years | 100 mcg of mRNA-1273: 56-70 Years | 25 mcg of mRNA-1273: 71+ Years | 50 mcg of mRNA-1273: 71+ Years | 100 mcg of mRNA-1273: 71+ Years
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 14/15 | 15/15 | 15/15 | 15/15 | 10/10 | 10/10 | 9/10 | 10/10 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mcg of mRNA-1273: 18-55 Years (N=15) | 50 mcg of mRNA-1273:18-55 Years (N=15) | 100 mcg of mRNA-1273: 18-55 Years (N=15) | 250 mcg of mRNA-1273: 18-55 Years (N=15) | 25 mcg of mRNA-1273: 56-70 Years (N=10) | 50 mcg of mRNA-1273: 56-70 Years (N=10) | 100 mcg of mRNA-1273: 56-70 Years (N=10) | 25 mcg of mRNA-1273: 71+ Years (N=10) | 50 mcg of mRNA-1273: 71+ Years (N=10) | 100 mcg of mRNA-1273: 71+ Years (N=10)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mcg of mRNA-1273: 18-55 Years (N=15) | 50 mcg of mRNA-1273:18-55 Years (N=15) | 100 mcg of mRNA-1273: 18-55 Years (N=15) | 250 mcg of mRNA-1273: 18-55 Years (N=15) | 25 mcg of mRNA-1273: 56-70 Years (N=10) | 50 mcg of mRNA-1273: 56-70 Years (N=10) | 100 mcg of mRNA-1273: 56-70 Years (N=10) | 25 mcg of mRNA-1273: 71+ Years (N=10) | 50 mcg of mRNA-1273: 71+ Years (N=10) | 100 mcg of mRNA-1273: 71+ Years (N=10)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scintillating scotoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotid duct obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral lichenoid reaction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site muscle weakness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exposure via inhalation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Smear cervix abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar II disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic spasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vasodilatation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 7 (7) | 4 (5) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 3 (3) | 12 (13) | 12 (14) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 5 (5)
Fatigue (General disorders) | 7 (9) | 10 (18) | 12 (16) | 10 (15) | 4 (6) | 5 (6) | 7 (10) | 3 (3) | 5 (9) | 7 (10)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 6 (6) | 8 (8) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaccination site erythema (General disorders) | 1 (1) | 4 (5) | 2 (4) | 4 (5) | 1 (2) | 1 (1) | 3 (3) | 3 (4) | 2 (2) | 4 (4)
Vaccination site induration (General disorders) | 0 (0) | 3 (3) | 3 (4) | 4 (7) | 5 (6) | 3 (3) | 3 (5) | 2 (2) | 2 (2) | 3 (3)
Vaccination site pain (General disorders) | 11 (20) | 14 (26) | 15 (29) | 15 (29) | 6 (8) | 9 (14) | 9 (16) | 8 (12) | 7 (11) | 10 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 2 (4) | 8 (8) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (8) | 8 (9) | 13 (17) | 6 (8) | 3 (3) | 7 (8) | 3 (4) | 2 (2) | 6 (8)
Headache (Nervous system disorders) | 4 (6) | 10 (13) | 10 (13) | 15 (21) | 3 (4) | 3 (4) | 7 (7) | 4 (5) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT04283461/Prot_002.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT04283461/SAP_001.pdf
  • Informed Consent Form (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT04283461/ICF_000.pdf